CLINICAL TRIAL: NCT03191695
Title: The Investigation of Necessity, Participation to Life of Children With Cerebral Palsy and Their Families
Brief Title: Participation to Life of Children With Cerebral Palsy
Acronym: PLCC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other); Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Mintaze Kerem Gunel, Prof. Dr., Hacettepe University
Other Study IDs: 116S359-1
Record Dates: First submitted 2017-06-16; First posted 2017-06-19 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Cerebral Palsy
Keywords: Participation; Activity; Cerebral Palsy; LIFE Habits (life-H); Gross Motor Function; Health-related Quality of Life; Family
MeSH Terms: conditions — Cerebral Palsy; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment via questionnaire — All the children will be assessed via assessment questionnaires.

SUMMARY:
Cerebral Palsy (CP) defined as a group of permanent impairments that is originating from non-progressive disorders that develop in the immature brain. CP leads activity limitations of movement and posture development. Motor problems in CP are usually accompanied by sensory and perceptual disorders, cognitive disorders, communication and behavioral disorders, epilepsy, and secondary musculoskeletal system problems. The first 20 years of life is characterized by rapid growth and specific changes in physical, social, and psychological development. Social participation and independence of children and youth are related to the changes in this period. Participation can be identified as being involved in life situations and it reflects the social aspect of functionality. The problems which can be come across in life situations are identified as participation limitation. In literature, no adequate study has investigated the functional inadequacy, activity and participation of children with CP; this project has been planned in order to specify the importance in rehabilitation interventions more detailed. This project aims to specify whether the functional levels correspond to the activity and participation limitations of children with CP living in Ankara city center and determine the effects of their functional status on activity, participation and quality of life. This investigation will be pioneer in indicating the activity and participation limitations of children with CP. According to the results, these limitations will be overcome and the quality of life of children with CP will be increased. The CP follow-up database in Ankara will be specified so their physical activity and participation levels will be followed periodically and CP profile will be determined in Ankara.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) defined as a group of permanent impairments that is originating from non-progressive disorders that develop in the immature brain. CP leads activity limitations of movement and posture development.The first 20 years of life is characterized by rapid growth and specific changes in physical, social, and psychological development. Social participation and independence of children and youth are related to the changes in this period. Participation can be identified as being involved in life situations and it reflects the social aspect of functionality. The problems which can be come across in life situations are identified as participation limitation. In the past, the impairment seen in child was concentrated and child was the passive receptor of treatment. Today, this view is changed and child is the active participant of the treatment of disability. The aim of treatment is identified as increasing the quality of life by supporting the activity and participation according to the priorities of the child and the parent.

In literature, no adequate study has investigated the functional inadequacy, activity and participation of children with CP; this project has been planned in order to specify the importance in rehabilitation interventions more detailed. This project aims to specify whether the functional levels correspond to the activity and participation limitations of children with CP living in Ankara city center and determine the effects of their functional status on activity, participation and quality of life. This investigation will be pioneer in indicating the activity and participation limitations of children with CP. According to the results, these limitations will be overcome and the quality of life of children with CP will be increased. The CP follow-up database in Ankara will be specified so their physical activity and participation levels will be followed periodically and CP profile will be determined in Ankara. Moreover, the results of this study will be shared with the Ministry of National Education, the Ministry of Family and Social Policies, and the Ministry of Health and this will bring a different viewpoint to the community-based rehabilitation services in Turkey. Furthermore, this study will be expected to motivate countrywide investigations.

In the project, Gross Motor Function Classification System (GMFCS) for the severity of the disability of people with CP, The Measure of Processes of Care (MPOC) for their care process, the Pediatric Outcomes Date Collection (PODCI) Instrument and Pediatric Quality of Life Questionnaire and The Child Health Quality (CHQ PF-50) for their health-related quality of life, the Manual Ability Classification System (MACS) for the manual abilities and the Communication Function Classification System (CFCS) for the communication skill and the Life Habits Questionnaire (LIFE-H) for the participation level and Impact on Family Scale (IPFAM) for family impact will be used and the outcomes will be analyzed by adequate statistical methods. It is intended to be discussed the findings of the project in national and international platforms.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed as cerebral palsy

Exclusion Criteria:

* Children whose family didn't accept to participate to study

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The subjects will be recruited from children who lives in Ankara city and, attend special education centers.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Life Habits Questionnaire (LIFE-H) | At baseline
  Assessing of the participation level of children

SECONDARY OUTCOMES:
Gross Motor Function Classification System (GMFCS) | At baseline
  Assessing severity of the disability of children
Pediatric Outcomes Date Collection (PODCI) (Questionnaire) | At baseline
  Assessing health-related quality of life of children by parent proxy questionnaire
Manual Ability Classification System (MACS) | At baseline
  Assessing the manual abilities
Communication Function Classification System (CFCS) | At baseline
  Assessing communication skill
The Child Health Quality (CHQ PF-50) | At baseline
  Assessing health-related quality of life
Pediatric Quality of Life Questionnaire (PedsQL) | At baseline
  Assessing health-related quality of life
The Measure of Processes of Care (MPOC) (Questionnaire) | At baseline
  Assessing health care process of children by parent proxy questionnaire
Impact on Family Scale (IPFAM) | At baseline
  Assessing family impact
Pediatric Evaluation of Disability Inventory | At baseline
  Assessing disability

CONTACTS AND LOCATIONS:
Overall Officials: Mintaze KEREM GÜNEL, Principal Investigator — Prof. Dr.
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Himuro N, Kozuka N, Mori M. Measurement of family-centred care: translation, adaptation and validation of the Measure of Processes of Care (MPOC-56 and -20) for use in Japan. Child Care Health Dev. 2013 May;39(3):358-65. doi: 10.1111/j.1365-2214.2012.01371.x. Epub 2012 Feb 28. PMID 22372945
- [Background] Bodkin AW, Robinson C, Perales FP. Reliability and validity of the gross motor function classification system for cerebral palsy. Pediatr Phys Ther. 2003 Winter;15(4):247-52. doi: 10.1097/01.PEP.0000096384.19136.02. PMID 17057460
- [Background] Berg M, Jahnsen R, Froslie KF, Hussain A. Reliability of the Pediatric Evaluation of Disability Inventory (PEDI). Phys Occup Ther Pediatr. 2004;24(3):61-77. doi: 10.1300/j006v24n03_05. PMID 15257969
- [Background] Damiano DL, Gilgannon MD, Abel MF. Responsiveness and uniqueness of the pediatric outcomes data collection instrument compared to the gross motor function measure for measuring orthopaedic and neurosurgical outcomes in cerebral palsy. J Pediatr Orthop. 2005 Sep-Oct;25(5):641-5. doi: 10.1097/01.bpo.0000167079.83835.22. PMID 16199947